CLINICAL TRIAL: NCT04258982
Title: The Copmparison of Accuracy of PtcCO2 and in PetCO2 in COPD Patients With NIV Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhenfeng He (Other)
Responsible Party: Sponsor-Investigator, Zhenfeng He, principal investigator, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: GIRH-201927
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AECOPD group: The study incruit AECOPD patients with type II respiratory failure who need the NIV treatment.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The chronic obstructive pulmonary disease (COPD) patients with type II respiratory failure always needs PaCO2 test to monitor the changes of disease. Method used mostly nowadays to detect PaCO2 is arterial puncture which is accurate but is invasive, painful and non-dynamic. Noninvasive measurement methods includes end-tidal CO2 (PetCO2), transcutaneous CO2 (PtcCO2) which can monitor the PaCO2 dynamically and noninvasively, but their accuracy is in controversy. Common PetCO2 is especially inaccurate in COPD patients while our team find that the accuracy can be improved by prolong expiration method (PetCO2 (P)).So the investigators want to compare the accuracy of PtcCO2 and PetCO2(P) in AECOPD patients during noninvasive ventilation(NIV).

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients with type II respiratory failure who need NIV treatment

Exclusion Criteria:

* hemodynamics is unstable;
* any other lung disease despite COPD;
* other diseases influencing experiments: Cognitive impairment disease mouth and nose trauma.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AECOPD patients with type II respiratory failure who need NIV treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
partial arterial pressure of end-tidal CO2 measured by prolong expiration method [PetCO2(P)] | 2 hours
  PetCO2(P) will be measured before and after NIV treatment.
partial arterial pressure of transcutaneous CO2 (PtcCO2) | 2 hours
  PtcCO2 will be measured before and after NIV treatment.
partial arterial pressure of carbon dioxide (PaCO2) | 2 hours
  PaCO2 will be measured before and after NIV treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided